CLINICAL TRIAL: NCT01688895
Title: Erythropoietic Protoporphyrias: Studies of the Natural History, Genotype-Phenotype Correlations, and Psychosocial Impact
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); Office of Rare Diseases (ORD) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 08-0959-04; HSM12-00307 (Other: Mount Sinai School of Medicine); U54DK083909 (NIH)
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Erythropoietic Protoporphyria; EPP; X-Linked Protoporphyria; XLP; XLPP; X-Linked Dominant Erythropoietic Protoporphyria; XLEPP; XLDP
Keywords: erythropoietic; protoporphyria; cutaneous; porphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Protoporphyria, Erythropoietic, X-Linked Dominant; Porphyrias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA extracted from peripheral blood sample or buccal (inside cheek) sampling for DNA analysis; whole blood in ACD anti-coagulant to establish a lymphoid cell line, red blood cells and plasma for biochemical assays.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Participants with Protoporphyrias: Individuals with a documented diagnosis of Erythropoietic Protoporphyria (EPP) or X-Linked Protoporphyria (XLP)

SUMMARY:
The initial objective of this protocol is to assemble a well-documented group of patients with confirmed diagnoses of the erythropoietic protoporphyrias, including autosomal recessive Erythropoietic Protoporphyria (EPP) and X-Linked Protoporphyria (XLP) for clinical, biochemical, and genetic studies. The long-term objectives are (1) to conduct a longitudinal investigation of the natural history, complications, and therapeutic outcomes in people with erythropoietic protoporphyria, (2) to systematically investigate the psychological effects of the erythropoietic protoporphyrias on children and adults, and (3) to investigate the correlation between the identified genotypes and the resulting clinical presentation, also determining the possible interaction of other genetic markers.

DETAILED DESCRIPTION:
The porphyrias are a group of rare metabolic diseases that may present in childhood or adult life and are due to deficiencies of enzymes in the heme biosynthetic pathway. The most common manifestations are related to accumulation of intermediates in the pathway and usually occur as acute neurological attacks (as in the acute or hepatic porphyrias), or cutaneous photosensitivity (as in the cutaneous porphyrias, including the erythropoietic protoporphyrias). Multiple mutations have been identified in each of the porphyrias. The risk of disability or death from these disorders is significant, in part because diagnosis is often delayed due to lack of adoption of diagnostic testing in clinical practice. Moreover, the natural history of these disorders is not well described and it is not known what determines differences in outcomes. New therapies are needed. For existing therapies, high-quality evidence on short and long term efficacy and safety is generally lacking. Therefore, the purpose of this study of a large group of patients with EPP and XLP is to provide a better understanding of the natural history of these disorders, as affected by available therapies, and to aid in developing new forms of treatment. Much of the data collected on subjects as participants in the Longitudinal Study of the Porphyrias will be accessed for this study specific to the investigation of the erythropoietic protoporphyrias. To maximize the information that can be informative in our objectives, additional data will be collected, including additional biochemical findings and EPP-specific psychosocial parameters.

The Office of Rare Diseases (ORD) of the National Institutes of Health (NIH) established a Rare Diseases Clinical Research Network (RDCRN) in collaboration with other NIH Institutes and currently has funded 19 rare diseases clinical research consortia and one Data Management and Coordinating Center. The Porphyrias Consortium was created as part of the RDCRN, to study the human porphyrias. The Porphyrias Consortium is a consortium of the academic institutions listed in the participating institutions table. All Centers in the Porphyrias Consortium are participating in this study. Additional centers may be added if funding is available.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must also be enrolled in the Longitudinal Study of the Porphyrias.
* Willing to sign informed consent form
* Biochemical findings - A marked increase in erythrocyte protoporphyrin [total erythrocyte protoporphyrin >200 ug/dL, or more than 1.5-fold increase (relative to ULN of 80 ug/dL)], with a predominance of free protoporphyrin (85-100% in EPP and 50-85% in XLP).
* Molecular findings - one of the following:

  1. A disease causing FECH mutation trans to the IVS3-48C>T low expression FECH allele
  2. Two disease-causing FECH mutations
  3. A gain-of-function ALAS-2 C-terminal deletion/exon 11 mutation (in XLP). If no mutation is found and subjects fulfill criteria 1-3 they are eligible for enrollment.

Exclusion Criteria:

* cases with elevations of porphyrins in urine, plasma or erythrocytes due to other diseases (i.e. secondary porphyrinuria or porphyrinemia), such as liver and bone marrow diseases [Gibson 2000].
* patients with a prior diagnosis of porphyria that cannot be documented by review of existing medical records or repeat biochemical or DNA testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the following resources:
  1. Patients followed by one of the Investigators
  2. The American Porphyria Foundation (APF)
  3. The Rare Diseases Clinical Research Network (RDCRN) Contact Registry
  4. Non-study Physician referrals
  5. Self-referrals, including family members of individuals diagnosed with Porphyria (proband) and other individuals who may have heard about the study from other subjects or prospective subjects.
  6. Medical Records Review
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-07; Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Balwani, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: Website for the Rare Diseases Clinical Research Network (RDCRN) Porphyrias Consortium (PC) — https://www.rarediseasesnetwork.org/cms/porphyrias

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Patients With EPP/XLP: Individuals with a documented diagnosis of Erythropoietic Protoporphyria (EPP) or X-Linked Protoporphyria (XLP)
Period: Overall Study
Arm/Group | Adult Patients With EPP/XLP
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Patients With EPP/XLP
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 2
Protoporphyria Type [Count of Participants; unit: Participants]
  Erythropoietic Protoporphyria - EPP | 143
  X-Linked Protoporphyria - XLP | 6
  Unknown type | 1
Age at Onset of Symptoms [Mean (Standard Deviation); unit: years] | 4.2 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: The Hospital Anxiety and Depression Scale (HADS)
Description: Questionnaire with 7 items for anxiety and 7 items for depression, each item is scored on a 4 point response 0 - 3, subscales 0-21, with full range from 0 to 42, with higher score indicating more severe anxiety or depression.
Time Frame: 1 weeks
Population: Data only for those who completed instrument included. A protocol modification to add the HADS tool was done after study initiation, therefore not all subjects received all tools.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Patients With EPP/XLP
Number analyzed (Participants) | 103
score on a scale
  Anxiety | 4.6 (4.1)
  Depression | 1.9 (2.1)

2. Primary Outcome: Illness Perception Questionnaire Revised (IPQR)
Description: Each item is scored on a likert scale from 1 (strongly disagree) to 5 (strongly agree). Items within each domain were totaled for final domain scores.
  Seven domains - Timeline (score 5-25), Consequences (score 6-30), Personal Control (score 6-30), Treatment Control (score 3-15), Illness Coherence (score 5-25), Timeline-Cyclical (score 4-20), and Emotional Representations (score 6-30). A modified version without the identity component was used as it was not applicable in EPP.
  Higher scores domains indicate overall strong beliefs that the disease is chronic and has a negative impact.
Time Frame: 1 week
Population: Data only for those who completed instrument included. A protocol modification to add the IPQR tool was done after study initiation, therefore not all subjects received all tools.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Patients With EPP/XLP
Number analyzed (Participants) | 104
score on a scale
  Timeline | 23.4 (2.2)
  Consequences | 23.2 (4.3)
  Personal Control | 19.0 (4.9)
  Treatment Control | 9.2 (2.8)
  Illness Coherence | 19.0 (4.2)
  Timeline - Cyclical | 10.5 (3.8)
  Emotional Representations | 18.8 (5.5)

3. Primary Outcome: EPP-Specific Tool
Description: Each item was scored from 0-3 on a Likert scale. There are 2 domains: S=disease severity and Q=QoL. Total scale for each domain transferred to 0-100 scale. Higher scores for the S domain reflect lower severity, and higher satisfaction/QoL for the Q domain. Total Score from 0-100, with higher score indicating higher quality of life.
Time Frame: 1 week
Population: Data only for those who completed instrument included. A protocol modification to add the EPP-Specific tool was done after study initiation, therefore not all subjects received all tools.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adult Patients With EPP/XLP
Number analyzed (Participants) | 107
units on a scale
  S Domain | 58.9 (30.8)
  Q Domain | 30.8 (27.4)
  Total Score | 54.3 (30.0)

4. Secondary Outcome: Sleep Disturbance PROMIS Scores
Description: Sleep Subscales: Pain Interference, Depression, Physical Function, Fatigue, Anxiety, Sleep Disturbance, Satisfaction with Social Roles, each subscale scored from 0-100 with higher score indicating more symptoms affecting sleep.
Time Frame: baseline
Population: *Only those subjects who completed the PROMIS was included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Patients With EPP/XLP
Number analyzed (Participants) | 117
score on a scale
  Pain Interference | 49.1 (9.7)
  Depression | 44.1 (8.4)
  Physical Function: number analyzed (Participants) | 116
  Physical Function | 52.5 (7.8)
  Fatigue | 46.6 (10.6)
  Anxiety: number analyzed (Participants) | 116
  Anxiety | 47.3 (10.0)
  Sleep Disturbance | 48.7 (8.9)
  Satisfaction with Social Roles | 54.9 (9.3)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Adult Patients With EPP/XLP
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT01688895/Prot_SAP_000.pdf